CLINICAL TRIAL: NCT05257109
Title: Water Content In E-Liquids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2000031495; 2U54DA036151-06 (NIH)
Record Dates: First submitted 2022-02-11; First posted 2022-02-25 (Actual); Results first posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: Nicotine E-Cigarette Use

STUDY DESIGN:
Intervention Model Description: Within subject design, all participants will receive all e-liquid flavors/water concentrations
Who Masked: Participant, Investigator
Masking Description: Double blind, both participant and investigator will be blind to e-liquid being administered
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental E-Liquid Order "A" (Experimental): All participants will be given all e-liquids (i.e. all 16 flavor*water concentration combinations (4 flavors and four water concentrations)) in this within subject cross-over design study. Participants will be randomized in the order in which they receive the flavor conditions (across the 2 visits). For each flavor condition, water order will be randomized.
  Interventions: Other: Water Concentration 1; Other: Water Concentration 2; Other: Water Concentration 3; Other: Water Concentration 4
- Experimental E-Liquid Order "B" (Experimental): All participants will be given all e-liquids (i.e. all 16 flavor*water concentration combinations (4 flavors and four water concentrations)) in this within subject cross-over design study. Participants will be randomized in the order in which they receive the flavor conditions (across the 2 visits). For each flavor condition, water order will be randomized.
  Interventions: Other: Water Concentration 1; Other: Water Concentration 2; Other: Water Concentration 3; Other: Water Concentration 4
- Experimental E-Liquid Order "C" (Experimental): All participants will be given all e-liquids (i.e. all 16 flavor*water concentration combinations (4 flavors and four water concentrations)) in this within subject cross-over design study. Participants will be randomized in the order in which they receive the flavor conditions (across the 2 visits). For each flavor condition, water order will be randomized.
  Interventions: Other: Water Concentration 1; Other: Water Concentration 2; Other: Water Concentration 3; Other: Water Concentration 4
- Experimental E-Liquid Order "D" (Experimental): All participants will be given all e-liquids (i.e. all 16 flavor*water concentration combinations (4 flavors and four water concentrations)) in this within subject cross-over design study. Participants will be randomized in the order in which they receive the flavor conditions (across the 2 visits). For each flavor condition, water order will be randomized.
  Interventions: Other: Water Concentration 1; Other: Water Concentration 2; Other: Water Concentration 3; Other: Water Concentration 4

INTERVENTIONS:
Other: Water Concentration 1 — E-liquid containing 36mg/ml pronated nicotine will be administered with no alteration to water concentration.
Other: Water Concentration 2 — E-liquid containing 36mg/ml pronated nicotine will be administered with 5% total water concentration of e-liquid.
Other: Water Concentration 3 — E-liquid containing 36mg/ml pronated nicotine will be administered with 10% total water concentration of e-liquid.
Other: Water Concentration 4 — E-liquid containing 36mg/ml pronated nicotine will be administered with 20% total water concentration of e-liquid.

SUMMARY:
This study looks at the effect of manipulating the water concentration of certain e-liquids on sensory perception.

DETAILED DESCRIPTION:
This study looks at the effect of manipulating water concentration on e-cigarettes that contain aldehyde flavor chemicals on sensory perception. Regular e-cigarette users will be asked to complete 2 lab sessions in which they will sample 4 nicotine containing e-liquids. Each e-liquid will be sampled in four water concentration manipulations. Researchers will examine influence of flavor and water concentrations on sensory experience including appeal/liking and irritation and harshness.

ELIGIBILITY:
Inclusion Criteria:

* at least 21 years old
* able to read/write
* >/= 6 mths e-cig use
* regular e-cig use (>/= 4 days/week)
* use of flavored e-cigs
* use of nicotine containing e-cigs
* urine cotinine >/= 200ng/ml
* no plan to quit e-cig use

Exclusion Criteria:

* breastfeeding, pregnant, trying to become pregnant
* Medical conditions that increase risk of respiratory problems among participants
* Current use of illegal substances
* Medical conditions increasing risk of respiratory problems in nonpatient populations
* Current diagnosis of an untreated psychiatric condition
* Not fully vaccinated for Coronavirus-19

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Davis, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 108 people were phone screened for eligibility. 54 attended an in person intake appointment. Of those, 31 met inclusion criteria and were enrolled in the study and 30 participants complete all study procedures.
Pre-assignment Details: 31 of 54 intakes were randomized to receive study procedures. 22 people did not meet inclusion criteria at the time of intake and were not enrolled and 1 person was not available at the time of the lab sessions to participate.
Groups:
- Experimental E-Liquid Order "A"; Experimental E-Liquid Order "B"; Experimental E-Liquid Order "C"; Experimental E-Liquid Order "D": All participants will be given all e-liquids (i.e. all 16 flavor*water concentration combinations (4 flavors and four water concentrations)) in this within subject cross-over design study. Participants will be randomized in the order in which they receive the flavor conditions (across the 2 visits). For each flavor condition, water will be presented in the same order from hypothesized least irritating to most irritating.
  Water Concentration 1: E-liquid containing 36mg/ml pronated nicotine will be administered with no alteration to water concentration.
  Water Concentration 2: E-liquid containing 36mg/ml pronated nicotine will be administered with 5% total water concentration of e-liquid.
  Water Concentration 3: E-liquid containing 36mg/ml pronated nicotine will be administered with 10% total water concentration of e-liquid.
  Water Concentration 4: E-liquid containing 36mg/ml pronated nicotine will be administered with 20% total water concentration of e-liquid.
Period: Overall Study
Arm/Group | Experimental E-Liquid Order "A" | Experimental E-Liquid Order "B" | Experimental E-Liquid Order "C" | Experimental E-Liquid Order "D"
Started | 10 | 8 | 6 | 7
Completed | 9 | 8 | 6 | 7
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental Order A-D (All Participants Received All Conditions, Order Was Randomized): All participants received all conditions, order was randomized
Arm/Group | Experimental Order A-D (All Participants Received All Conditions, Order Was Randomized)
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 18
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Irritation/Harshness
Description: Change in irritation at each water level as measured by the computerized Generalized Labeled Magnitude Scale (gLMS). Participants will self-report their responses using a computer mouse to indicate where on the scale response falls. The Generalized Labeled Magnitude Scales (gLMS) are category ratio scales with seven semantic labels: "no sensation", "barely detectable", "weak", "moderate", "strong", "very strong", and "strongest imaginable", positioned quasi-logarithmically as per empirically determined semantic magnitudes on a 0-100 scale (strongest imaginable at the 100 end).
Time Frame: immediately after intervention, up to 15 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- No Water Added: All participants received all conditions, order was randomized
- 5% Water Added; 10% Water Added; 20% Water Added: All participants received all conditions
Arm/Group | No Water Added | 5% Water Added | 10% Water Added | 20% Water Added
Number analyzed (Participants) | 31 | 31 | 31 | 31
units on a scale | 1.04 (.05) | 1.07 (.05) | 1.03 (.05) | 1.01 (.05)
Statistical Analysis 1: Comparison: No Water Added vs 5% Water Added vs 10% Water Added vs 20% Water Added; Test type: Other — Mixed effects models with water concentration as the within subject factor and irritation as outcome. Outcome analyses will be intent-to-treat and using mixed-effects models. If model assumptions will appear to be violated, we will transform the data or fit more flexible generalized linear or nonparametric mixed models. A significant main effect of condition will be considered supportive of our hypothesis. Formal power analyses were not conducted for this pilot study; p = 0.0014, Mixed Models Analysis — Significant p-value set at <0.05; Median Difference (Final Values) = 0.67

2. Primary Outcome: Appeal Assessed Using the Labeled Hedonic Scale (LHS) Ranging From -100 to 100
Description: Change in appeal at each water level as measured by the computerized Labeled Hedonic Scale (LHS). Participants will self-report their responses using a computer mouse to indicate where on the scale response falls. The Labeled Hedonic Scale (LHS) is a bipolar category ratio scale that ranges from -100 (most disliked, minimum score) to 100 (most liked, maximum score), with 'neither liked nor disliked' as midpoint (0). Scores range from -100 (minimum) to 100 (maximum). Negative scores indicate dislike (lack of appeal) and positive scores indicate liking (appeal).
Time Frame: immediately after intervention, up to 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale (-100 to 100)
Arm/Group | No Water Added | 5% Water Added | 10% Water Added | 20% Water Added
Number analyzed (Participants) | 31 | 31 | 31 | 31
score on a scale (-100 to 100) | 9.91 (3.78) | 10.41 (3.79) | 7.1 (3.79) | 3.87 (3.79)
Statistical Analysis 1: Comparison: No Water Added vs 5% Water Added vs 10% Water Added vs 20% Water Added; Test type: Other — Mixed effects models with water concentration as the within subject factor and LHS as outcome. Outcome analyses will be intent-to-treat and using mixed-effects models. If model assumptions will appear to be violated, we will transform the data or fit more flexible generalized linear or nonparametric mixed models. A significant main effect of condition will be considered supportive of our hypothesis. Formal power analyses were not conducted for this pilot study; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = 1.55

3. Primary Outcome: Appeal Assessed Using the Drug Effects Questionnaire (DEQ)
Description: Change in appeal at each water level as measured by the computerized version of the Drug Effects Questionnaire (DEQ). Participants will self-report their responses using a computer mouse to indicate where on the scale response falls. A modified version of the Drug Effects Questionnaire (DEQ) will be used in which participants rate acute responses to the e-cigarette on a 0-100mm scale from "not at all" (0mm) to "extremely" (100mm).
Time Frame: immediately after intervention, up to 15 minutes
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | No Water Added | 5% Water Added | 10% Water Added | 20% Water Added
Number analyzed (Participants) | 31 | 31 | 31 | 31
score on a scale | 48.99 (3.71) | 47.94 (3.71) | 45.94 (3.71) | 42.97 (3.72)
Statistical Analysis 1: Comparison: No Water Added vs 5% Water Added vs 10% Water Added vs 20% Water Added; Test type: Other — Mixed effects models with water concentration as the within subject factor and DEQ as outcome. Outcome analyses will be intent-to-treat and using mixed-effects models. If model assumptions will appear to be violated, we will transform the data or fit more flexible generalized linear or nonparametric mixed models. A significant main effect of condition will be considered supportive of our hypothesis. Formal power analyses were not conducted for this pilot study; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = 3.28

ADVERSE EVENTS:
Time Frame: Data was collected from August 2022 to March 2023 and adverse events were assessed during that time. Participants were monitored for adverse events during the duration of their participation (i.e. they were asked about adverse events and monitored for AEs during Labs 1 and 2). For each participant the time they were enrolled varied, but it was approximately 1-2 weeks.
Description: Does not differ from clinical trials definition
Groups:
- Experimental Order A; Experimental Order B; Experimental Order C; Experimental Order D: All participants will be given all e-liquids (i.e. all 16 flavor*water concentration combinations (4 flavors and four water concentrations)) in this within subject cross-over design study. Participants will be randomized in the order in which they receive the flavor conditions (across the 2 visits). For each flavor condition, water will be presented in the same order from hypothesized least irritating to most irritating.
  Water Concentration 1: E-liquid containing 36mg/ml pronated nicotine will be administered with no alteration to water concentration.
  Water Concentration 2: E-liquid containing 36mg/ml pronated nicotine will be administered with 5% total water concentration of e-liquid.
  Water Concentration 3: E-liquid containing 36mg/ml pronated nicotine will be administered with 10% total water concentration of e-liquid.
  Water Concentration 4: E-liquid containing 36mg/ml pronated nicotine will be administered with 20% total water concentration of e-liquid.
Arm/Group | Experimental Order A | Experimental Order B | Experimental Order C | Experimental Order D
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/6 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT05257109/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT05257109/ICF_002.pdf